CLINICAL TRIAL: NCT02347839
Title: A Multicenter Phase II Trial of Neoadjuvant Gefitinib Followed by Surgery, Followed by Adjuvant Gefitinib in Patients With Unresectable Stage III Non-Small Cell Lung Cancer Harboring Activating Epidermal Growth Factor Receptor Mutations.
Brief Title: NEoadjuvant Gefitinib fOllowed by Surgery and gefiTinib In unresectAble sTage III NSCLC With EGFR Mutations.
Acronym: NEGOTIATE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1004; wsy005 (Other: Guangdong Province Association Study of Thoracic Oncology)
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental): Gefitinib-surgery-gefitinib. Induction gefitinib therapy was given for 8 weeks. Patients' resectability was assessed after 8-week gefitinib. Adjuvant gefitinib was given within 3-6 weeks after surgery until progression or unacceptable toxic effects.
  Interventions: Procedure: Gefitinib-surgery-gefitinib

INTERVENTIONS:
Procedure: Gefitinib-surgery-gefitinib — neoadjuvant gefitinib followed by surgery, followed by adjuvant gefitinib
  Other Names: neooadjuvant gefitinib followed by surgery and gefitinib

SUMMARY:
The purpose of this study is to studying neoadjuvant gefitinib followed by surgery, followed by adjuvant gefitinib to see how well it works in treating patients with unresectable stage III NSCLC harboring EGFR mutations.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the recommended therapeutic approach for patients with unresectable stage III non-small cell lung cancer (NSCLC), although surgery offers the chance of cure. With combined-modality therapy with radiation therapy and chemotherapy, the prognosis of stage III NSCLC remains poor. Gefitinib has shown great efficacy in NSCLC patients with EGFR mutations. This study is to studying neoadjuvant gefitinib followed by surgery, followed by adjuvant gefitinib to see how well it works in treating patients with unresectable EGFR mutant stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Target population is unresectable stage III (III A-bulky N2, III B) NSCLC with EGFR activating mutation in exon 19 or 21
* Written informed consent provided
* Aged 18-75 years
* Able to comply with the required protocol and follow-up procedures
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Had a life expectancy of 12 weeks or more
* Adequate hematological function, liver function and renal function
* Female participants should not be pregnant or breast-feeding

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of this product
* Inability to comply with protocol or study procedures
* Had had previous chemotherapy, radiotherapy, or agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab)
* Had a history another malignancy in the last 5 years with the exception of cured basal cell carcinoma of the skin, cured in situ carcinoma of the uterine cervix and cured epithelial carcinoma of the bladder
* Interstitial pneumonia
* Eye inflammation not fully controlled or conditions predisposing the subject to this
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease)
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast-feeding women
* History of neurologic or psychiatric disorders
* Ingredients mixed with small cell lung cancer patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01; Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | 3 months

SECONDARY OUTCOMES:
Number of participants with perioperative complications | 1 year
Event-free survival | 2 years after the last patient is randomized
  Event-free survival was assessed from randomization to disease recurrence/progression or death from any cause.
Overall survival | 2 years after the last patient is randomized
  Overall survival was assessed from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, Principal Investigator — Guangdong Province Association Study of Thoracic Oncology
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China